CLINICAL TRIAL: NCT05714904
Title: An Exploratory Clinical Study on Single Subretinal Injection of ZVS101e (rAAV2/8-hCYP4V2) Into Eyes With Bietti's Crystalline Dystrophy (BCD)
Brief Title: Safety and Tolerability of ZVS101e in Patients With Bietti 's Crystalline Dystrophy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZVS101e-01
Record Dates: First submitted 2022-12-13; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Bietti's Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): 2 cohorts of 3 patients each. All the patients enrolled in the study will receive a single subretinal injection in one eye.
  Cohort 1: Subretinal administration of a single low dose ZVS101e at Day 0. Cohort 2: Subretinal administration of a single high dose ZVS101e at Day 0.
  Interventions: Drug: ZVS101e

INTERVENTIONS:
Drug: ZVS101e — ZVS101e is developed by Chigenovo Co., Ltd., it contains recombinant adeno-associated virus serotype 8 (rAAV8) vectors which carry human CYP4V2 gene.
  Other Names: rAAV2/8-hCYP4V2; rAAV8-hCYP4V2

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of an adeno-associated virus vector expressing CYP4V2 in patients with Bietti's crystalline dystrophy (BCD).

DETAILED DESCRIPTION:
This is a single-arm, open-label, and single-center study of ZVS101e in patients with BCD. A total of 6 participants will be enrolled. A retinal surgeon will administer the vector by subretinal injection. Safety, efficacy and vector shedding characteristics of ZVS101e are then measured over 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to adhere to protocol as evidenced by written informed consent;
2. Patients with clinical diagnosis of Bietti's crystalline dystrophy (BCD) (age ≥ 18 years) (the age is based on the time of signing the informed consent form);
3. Genetic test confirmed to carry two pathogenic variants of CYP4V2 and carry no pathogenic mutations of other ophthalmic genetic diseases;
4. Agree to use reliable barrier contraception for 2 year after administration of ZVS101e;
5. The study eye must meet the following requirements: BCVA between 2.3 LogMAR and 0.5 LogMAR (including 2.3 LogMAR and 0.5 LogMAR); No refractive medium turbidity that affects fundus examination; Visible photoreceptor (outer nuclear) layer on a standard optical coherence tomography (OCT) scan.

Exclusion Criteria:

1. Lack of sufficient viable retinal cell. Specifically, if indirect ophthalmoscopy reveals less than I disc area of retina which is not involved by complete retinal degeneration, these eyes will be excluded. In addition, in eyes where OCT scans of sufficient quality can be obtained, areas of retina with thickness measurements less than 100 μm, or absence of neural retina, will not be targeted for delivery of AAV2-hCYP4V2;
2. Existing or pre-existing of choroidal neovascular (CNV) lesions that were secondary to BCD, or other eye conditions interfering with the surgery or the interpretation of the clinical endpoint, in the investigators' opinion;
3. The study eye has been treated with other drugs within 3 months that could affect the evaluation of the investigational drug (such as ranibizumab, bevacizumab, aflibercept, conbercept);
4. The study eye has been treated with the following intraocular procedures: retinal detachment surgery, vitrectomy;
5. Pre-existing eye conditions that the investigator evaluates could interfere with ocular evaluation, preclude surgery, interfere with interpretation of study endpoints or surgical complications (such as glaucoma, high refractive error, diabetes retinopathy or retinal vasculitis );
6. Currently taking or may require systemic medications that can cause ocular toxicity, such as psoralen, risedronate, or tamoxifen;
7. Patient with allergic constitution (such as those allergic to two or more drugs and food);
8. Those with the following laboratory abnormalities which are clinically significant:

   Liver function: chronic liver disease, ALT increased >3 times the upper limit of normal; With uncontrolled hypertension, mean systolic blood pressure ≥ 160 mmHg or mean diastolic blood pressure ≥ 100 mmHg; With uncontrolled diabetes, HbA1c>10%; Patients with abnormal coagulation function (prothrombin time ≥ upper limit of normal (3 seconds' longer), activated partial thromboplastin time ≥ upper limit of normal (10 seconds' longer)); Serum virology test: Active hepatitis B, hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) or syphilis antibody positive; Abnormality of tumor markers (alpha fetoprotein, carcinoembryonic antigen, CA125 carbohydrate antigen, CA153 carbohydrate antigen, CA199 carbohydrate antigen)
9. Having any past or present medical history that may affect the safety of the trial or the in vivo process of the drug, especially the medical history of cardiovascular, hepatic, renal, endocrine, gastrointestinal, pulmonary, neurological, hematological, oncologic, immunological or metabolic disorders and others that are thought clinically significant by the investigator, such as diabetes, severe cardiac failure (New York Heart Association Class III and IV);
10. Participation in any medicine or medical device clinical trials within 3 months prior to enrollment;
11. Neutralizing antibodies to rAAV> 1:1000 by immunologic test;
12. For females in pregnancy or lactation period;
13. Any other conditions which leads the investigator to determine the participant is unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and systemic adverse events (AEs) after ZVS101e treatment. | Baseline up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of ocular and systemic serious adverse events (SAEs) after ZVS101e treatment. | Baseline up to Week 52
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following:
  Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Type and severity of ocular and systemic AEs and SAEs after ZVS101e treatment. | Baseline up to Week 52
  Safety as the primary endpoint will be assessed by best-corrected visual acuity (BCVA), slit-lamp examination, ophthalmoscopy, fundus photography, intraocular pressure (IOP), optical coherence tomography (OCT), laboratory tests, vital signs, physical examinations, electrocardiogram (ECG), immunopathology and biodistribution of ZVS101e.

SECONDARY OUTCOMES:
Mean change from baseline in BCVA after ZVS101e treatment; | Baseline up to Week 52
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart.
Change from Baseline in visual field | Baseline up to Week 52
  Visual field will be assessed by Humphrey perimetry.
Change from Baseline in contrast sensitivity | Baseline up to Week 52
  Change from baseline in contrast sensitivity will be measured using the CSV-1000E instrument.
Change from Baseline in color vision | Baseline up to Week 52
  Subjects' color vision was classified and graded by having them identify the pictures within Color Vision Examination Plates.
Change from Baseline in retinal thickness | Baseline up to Week 52
  Retinal thickness will be assessed for both eyes using OCT.
Change from Baseline in NEI VFQ-25 total score | Baseline up to Week 52
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.
Change from Baseline in multi-luminance mobility test (MLMT) | Baseline up to Week 52
  MLMT was assessed using both eyes at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night).
Change from Baseline in fundus autofluorescence (FAF). | Baseline up to Week 52
  FAF is a noninvasive test to explore the health and metabolic status of retinal pigment epithelial cell/photoreceptor complex.
Change from Baseline in mfERG | Baseline up to Week 52
  The measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV).
Incidence of ocular and systemic AEs after ZVS101e treatment. | Week 53 to Week 104
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of ocular and systemic SAEs after ZVS101e treatment. | Week 53 to Week 104
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following:
  Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Type and severity of ocular and systemic AEs and SAEs after ZVS101e treatment. | Week 53 to Week 104
  Safety will be assessed by best-corrected visual acuity (BCVA), slit-lamp examination, ophthalmoscopy, fundus photography, intraocular pressure (IOP), optical coherence tomography (OCT), laboratory tests, vital signs, physical examinations, electrocardiogram (ECG), immunopathology and biodistribution of ZVS101e.

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Dou, MD, Principal Investigator — Peking University
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia R, Meng X, Chen S, Zhang F, Du J, Liu X, Yang L. AAV-mediated gene-replacement therapy restores viability of BCD patient iPSC derived RPE cells and vision of Cyp4v3 knockout mice. Hum Mol Genet. 2023 Jan 1;32(1):122-138. doi: 10.1093/hmg/ddac181. PMID 35925866